CLINICAL TRIAL: NCT06828432
Title: Validation of Three Non-invasive Hemodynamic Monitoring Systems for Determining Measures of Volume Responsiveness, Ventriculo-arterial Coupling and Cardiac Output
Brief Title: CTICU Device Study CRUISE
Acronym: CRUISE
Status: Enrolling by invitation | Type: Observational
Sponsor: Hernando Gomez (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Hernando Gomez, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY24080125; HT9425-24-C-0121 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2025-01-13; First posted 2025-02-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Open Heart Surgery
Keywords: Heart, Surgery, ICU, Monitor, Blood Pressure, Measurement; non-invasive; responsiveness; cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CRUISE CTICU CareTaker Vitalstream Device — The CareTaker Vitalstream device is a patented PDA technology and artificial intelligence algorithms derive continuous hemodynamic parameters by analyzing reflective pulse wave analyzes the pulse pressure waveform at 500 times per second, isolates the individual central aortic pulses that give rise to the observed pulse shape, reads central aortic measurements therefore eliminating the effects of hydrostatic pressure, and tracks vascular tone.
Device: CRUISE CTICU CNAP Device — The CNAP Monitor provides advanced hemodynamic information from the non-invasive reusable CNAP finger sensor. It supports your Goal Directed Therapy whenever an arterial line is not indicated. Patient-friendly, easy-to-use, cost-efficient. CNAP Monitor offers a unique set of parameters to support your daily routine - all non-invasive & continuous allowing for perioperative fluid management even in low and moderate-risk surgeries and patients.
Device: CRUISE CTICU Edwards Clearsight Device — The Edwards ClearSight system provides continuous blood pressure and advanced hemodynamic parameters from a noninvasive finger cuff. Continuous data offered by the ClearSight system enables you to proactively optimize perfusion through hemodynamic management.

SUMMARY:
The goal of this study evaluate three novel, Food and Drug Administration (FDA)-approved devices currently used to monitor blood pressure and the amount of blood that the heart pumps during each beat.

These devices are the ClearSight (Edwards Life Sciences), CareTaker (CareTaker Medical) and CNAP (CNS Systems). These devices measure blood pressure, how much blood the heart is pumping around the body each minute and on a heartbeat to heartbeat basis and other parameters that can tell the doctor if the patient will benefit from specific treatments. The purpose of this study is to determine the accuracy of these devices. This knowledge will help us understand how investigators can use such non-invasive devices to care for patients at less risk than the devices currently used for such purposes.

The main question the study aims to answer is:

• What monitor is the most accurate in capturing non-invasive patient data?

DETAILED DESCRIPTION:
Investigators will compare predictors of preload responsiveness, including pulse pressure variation (PPV) and stroke volume variation (SVV), and arterial dynamic elastance (Eadyn) in all patients and estimates of cardiac output (CO) in patients with an indwelling pulmonary artery catheter. in 50 intensive care unit, intubated patients during the patient's normal course of treatment using their usually present invasive monitoring devices for the first 8 hours following cardiac surgery.

The primary goal of the study will be to compare PPV, SVV and Eadyn measured by the non-invasive monitors ClearSight, CareTaker and CNAP versus a reference standard that uses invasive arterial pressure waveform data, which in this case will be the LiDCO monitor & FloTrac monitor. Investigators will calculate accuracy, precision and concordance of each of the parameters measured during steady state conditions and after specific interventions including the administration of crystalloid fluid boluses and changes in vasoactive or inotropic medications. As a secondary objective, investigators will compare measures of CO by the same non-invasive monitors with the pulmonary artery catheter as a reference standard during the same conditions as above (i.e., steady state conditions, and before/after interventions). CO will therefore be only compared in patients that have a pulmonary artery catheter in place.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Male and female patients following cardiac surgery admitted to the CTICU with or without a pulmonary artery catheter

Exclusion Criteria:

* Subjects whose sternum remains open post-surgery and/or the presence of a LV ventricular assist device.
* Presence of a any ventricular assist device, ECMO, Impella, durable LVAD, or central L/RVAD.
* Spontaneous breathing activity upon coming out of the operating room (i.e., patients extubated in the operating room).
* Presenting chronic atrial fibrillation, refractory acute atrial fibrillation to medical therapy or frequent extra-systoles.
* Children will be excluded from this study. The hospital unit where all subjects will be recruited is for adults' (ages 18 and up) only. Gender, racial and ethnic sub groups will not be explicitly excluded.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with estimates of cardiac output (CO) in patients with an indwelling pulmonary artery catheter. in 50 intensive care unit, intubated patients during the patient's normal course of treatment using their usually present invasive monitoring devices for the first 8 hours following cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Stroke Volume Variation | 8 hours
  The Stroke Volume Variation (SSV) will be collected continuously for 8 hours using all 3 devices (ClearSight, CareTaker and CNAP). The metric of performance will be the precision, accuracy and concordance assessed using Bland Altman analysis and Pearson's moment analysis comparing SVV from each of the non-invasive monitors with the reference standard obtained from the analysis of the arterial pressure waveform. Measurement of SVV, PPV, Eadyn and CO from non-invasive monitors will be obtained continuously, but the quantity will be recorded at different timepoints including: Baseline, every 30 min after baseline, before each bolus of crystalloid fluid or blood product (within 5 minutes of administration, after each bolus of crystalloid fluid or blood product (within 5 minutes of stopping), before each change in vasopressors or inotropes (within 5 minutes of administration), after each change in vasopressors or inotropes (within 5 minutes of stopping), before changing ventilatory mode.
Pulse Pressure Variation (PPV) | 8 hours
  The Pulse Pressure Variation will be collected continuously for 8 hours using all 3 devices (ClearSight, CareTaker and CNAP). The metric of performance will be the precision, accuracy and concordance assessed using Bland Altman analysis and Pearson's moment analysis comparing PPV from each of the non-invasive monitors with the reference standard obtained from the analysis of the arterial pressure waveform. This metric of performance will be reported. The most reliable device will be based on the metric of performance - that is, the most precise, accurate and concordant. Measurement of SVV, PPV, Eadyn and CO from non-invasive monitors will be obtained continuously, but the quantity will be recorded at different timepoints including: Baseline, every 30 min after baseline, before each bolus of crystalloid fluid or blood product (within 5 minutes of administration, after each bolus of crystalloid fluid or blood product (within 5 minutes of stopping), before each change in vasopressors.
Arterial Dynamic Elastance (Eadyn) | 8 hours
  The Arterial Dynamic Elastance (Eadyn) will be collected continuously for 8 hours using all 3 devices (ClearSight, CareTaker and CNAP). The metric of performance will be the precision, accuracy and concordance assessed using Bland Altman analysis and Pearson's moment analysis comparing Eadyn from each of the non-invasive monitors with the reference standard obtained from the analysis of the arterial pressure waveform. This metric of performance will be reported. The most reliable device will be based on the metric of performance - that is, the most precise, accurate and concordant. Measurement of SVV, PPV, Eadyn and CO from non-invasive monitors will be obtained continuously, but the quantity will be recorded at different timepoints including: Baseline, every 30 min after baseline, before each bolus of crystalloid fluid or blood product (within 5 minutes of administration, after each bolus of crystalloid fluid or blood product (within 5 minutes of stopping).

SECONDARY OUTCOMES:
Cardiac Output | 8 hours
  Compare measures of CO by the ClearSight, CareTaker and CNAP non-invasive monitors with the pulmonary artery catheter as a reference standard during the same conditions as above (i.e., steady state conditions, and before/after interventions). CO will therefore be only compared in patients that have a pulmonary artery catheter in place. Measurement of SVV, PPV, Eadyn and CO from non-invasive monitors will be obtained continuously, but the quantity will be recorded at different timepoints including: Baseline, every 30 min after baseline, before each bolus of crystalloid fluid or blood product (within 5 minutes of administration, after each bolus of crystalloid fluid or blood product (within 5 minutes of stopping), before each change in vasopressors or inotropes (within 5 minutes of administration), after each change in vasopressors or inotropes (within 5 minutes of stopping), before changing ventilatory mode to pressure support ventilation, after 30+/-5 minutes of changing ventilatory.
Volume Responsiveness Collection | 8 hours
  The performance of ClearSight, CareTaker and CNAP in predicting volume responsiveness as compared to LiDCO, using a change of 10% or more in CO in response to fluid administration measured with a PAC as the definition of volume responsiveness. Measurement of SVV, PPV, Eadyn and CO from non-invasive monitors will be obtained continuously, but the quantity will be recorded at different timepoints including: Baseline, every 30 min after baseline, before each bolus of crystalloid fluid or blood product (within 5 minutes of administration, after each bolus of crystalloid fluid or blood product (within 5 minutes of stopping), before each change in vasopressors or inotropes (within 5 minutes of administration), after each change in vasopressors or inotropes (within 5 minutes of stopping), before changing ventilatory mode to pressure support ventilation, after 30+/-5 minutes of changing ventilatory mode to pressure support ventilation, before extubation (within 5minutes), after extubation .

CONTACTS AND LOCATIONS:
Overall Officials: Hernando Gomez, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We will not share any data outside our study team. The DOD requires all vendors to sign NDAs and commit to the rules of the study. Any party that may have access to the data will be part of the study team and committed thru NDAs & subcontracts.

REFERENCES:
- [Background] Michard F, Chemla D, Richard C, Wysocki M, Pinsky MR, Lecarpentier Y, Teboul JL. Clinical use of respiratory changes in arterial pulse pressure to monitor the hemodynamic effects of PEEP. Am J Respir Crit Care Med. 1999 Mar;159(3):935-9. doi: 10.1164/ajrccm.159.3.9805077. PMID 10051276
- [Background] Ramsey SD, Saint S, Sullivan SD, Dey L, Kelley K, Bowdle A. Clinical and economic effects of pulmonary artery catheterization in nonemergent coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2000 Apr;14(2):113-8. doi: 10.1016/s1053-0770(00)90001-6. PMID 10794325